CLINICAL TRIAL: NCT00542269
Title: A Twelve Week, Randomized, Double-blind, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren/Ramipril/Amlodipine (300/10/5-10 mg) Compared to the Combinations of Ramipril/Amlodipine (10/5-10 mg) and Aliskiren/Amlodipine (300/5-10 mg) in Patients With Essential Hypertension and Metabolic Syndrome Not Adequately Responsive to Amlodipine 5-10 mg
Brief Title: Efficacy and Safety of Aliskiren/Ramipril/Amlodipine Compared With Ramipril/Amlodipine and Aliskiren/Amlodipine in Patients With Metabolic Syndrome
Acronym: ALTO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination of the study due to slow recruitment.
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100AGB01
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension With Metabolic Syndrome
Keywords: Hypertension; Metabolic Syndrome; Dual combination therapy; Triple combination therapy; Aliskiren; Direct Renin inhibitor
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Amlodipine; aliskiren; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aliskiren / ramipril / amlodipine (Experimental): 6 weeks treatment with aliskiren 150 mg tablets, ramipril 5 mg capsules, and amlodipine 5-10 mg tablets followed by an additional 6 weeks treatment with aliskiren 300 mg tablets, ramipril 10 mg capsules, and amlodipine 5-10 mg tablets. Patients received amlodipine 5 mg (or 10 mg if they were receiving 10 mg prior to study start). Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
  Interventions: Drug: Amlodipine; Drug: Aliskiren; Drug: Ramipril
- Aliskiren / amlodipine (Experimental): 6 weeks treatment with aliskiren 150 mg tablets, ramipril 5 mg placebo capsules, and amlodipine 5-10 mg tablets followed by an additional 6 weeks treatment with aliskiren 300 mg tablets, ramipril 10 mg placebo capsules, and amlodipine 5-10 mg tablets. Patients received amlodipine 5 mg (or 10 mg if they were receiving 10 mg prior to study start). Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
  Interventions: Drug: Amlodipine; Drug: Aliskiren
- Ramipril / amlodipine (Active Comparator): 6 weeks treatment with aliskiren 150 mg placebo tablets, ramipril 5 mg capsules, and amlodipine 5-10 mg tablets followed by an additional 6 weeks treatment with aliskiren 300 mg placebo tablets, ramipril 10 mg capsules, and amlodipine 5-10 mg tablets. Patients received amlodipine 5 mg (or 10 mg if they were receiving 10 mg prior to study start). Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
  Interventions: Drug: Amlodipine; Drug: Ramipril

INTERVENTIONS:
Drug: Amlodipine — amlodipine 5-10 mg tablets. Patients received amlodipine 5 mg (or 10 mg if they were receiving 10 mg prior to study start). Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
Drug: Aliskiren — aliskiren 150-300 mg tablets. Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
  Arms: Aliskiren / amlodipine; Aliskiren / ramipril / amlodipine
Drug: Ramipril — ramipril 5-10 mg capsules. Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
  Arms: Aliskiren / ramipril / amlodipine; Ramipril / amlodipine

SUMMARY:
This proof of concept study is designed to evaluate the efficacy and safety of the combination therapy of aliskiren and ramipril as add-on to amlodipine in the treatment of patients with essential hypertension and metabolic syndrome who do not respond adequately to amlodipine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18-75 years of age.
* Male or female patients are eligible.
* Patients with a diagnosis of hypertension:
* Newly diagnosed patients or patients who have not been treated for hypertension within the 4 weeks prior to Visit 1 must have a mean sitting systolic blood pressure (MSSBP) > 150 mmHg and < 180 mmHg at Visit 1.
* Patients treated with antihypertensive monotherapy must have a MSSBP ≥ 140 mmHg and <180 mmHg at Visit 1.
* Patients taking amlodipine monotherapy MSSBP > 140 mmHg and < 180 mmHg at visit 1.
* All patients must have a MSSBP ≥ 140 mmHg and < 180 mmHg at Visit 3, the end of the amlodipine run-in period.
* Metabolic syndrome.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written inform consent form).

Exclusion Criteria:

* Severe hypertension (office cuff MSDBP ≥ 115 mmHg and/or MSSBP ≥ 180 mmHg).
* History or evidence of a secondary form of hypertension.
* History of hypertensive encephalopathy or cerebrovascular accident, transient ischemic cerebral attack (TIA), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI).
* Serum sodium < 135 mmol/L at Visit 1 if confirmed on repeat sample.
* Serum potassium < 3.5 mmol/L or ≥ 5.3 mmol/L at Visit 1, if confirmed on repeat sample.
* Type 1 diabetes mellitus.
* Type 2 diabetes if oral hypoglycaemic therapy changed (dose change or medication change) in previous 3 months.
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Great Britian
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren /Amlodipine: 6 weeks treatment with aliskiren 150 mg tablets, ramipril 5 mg placebo capsules, and amlodipine 5-10 mg tablets followed by an additional 6 weeks treatment with aliskiren 300 mg tablets, ramipril 10 mg placebo capsules, and amlodipine 5-10 mg tablets. Patients received amlodipine 5 mg (or 10 mg if they were receiving 10 mg prior to study start). Each dose was to be taken orally with water once daily at approximately 8:00 A.M. with or without food, except on the morning of an office/clinic visit, when the study drug was to be taken at the site after the visit procedures had been completed.
Period: Overall Study
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine
Started | 61 | 60 | 57
Completed | 48 | 54 | 51
Not Completed | 13 | 6 | 6
Not completed — Adverse Event | 10 | 4 | 5
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Administrative problems | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine | Total
Number analyzed (Participants) | 61 | 60 | 57 | 178
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.90) | 58.3 (8.95) | 59.1 (8.86) | 59.6 (8.95)
Age, Customized [Number; unit: participants]
  < 65 years | 37 | 47 | 42 | 126
  ≥ 65 years | 24 | 13 | 15 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 19 | 54
  Male | 44 | 42 | 38 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study - Aliskiren/Ramipril/Amlodipine vs Ramipril/Amlodipine)
Description: Automated blood pressure determinations were made with the Omron HEM-705CP blood pressure monitor at trough (24 hours ± 3 hours post-dose) and recorded at all study visits following detailed directions specified in the study protocol. Three readings were made and msSBP was calculated as the average of the 3 readings. In the event of aberrant readings, ie, the lowest reading was ≥ 10 mmHg systolic or ≥ 5 mmHg diastolic lower than the highest of the 3 readings, 3 additional readings were obtained. A negative change indicates improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Ramipril / Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 61 | 57
mmHg | -12.8 (1.56) | -10.9 (1.59)

2. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study - Aliskiren/Amlodipine vs Ramipril/Amlodipine
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: Intent-to-treat (ITT) population. All patients that received at least 1 dose of study drug and had baseline and at least 1 post-baseline assessment of the variable.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 60 | 57
mmHg | -12.4 (1.36) | -10.0 (1.39)

3. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study - Aliskiren/Ramipril/Amlodipine vs Ramipril/Amlodipine
Description: Automated blood pressure determinations were made with the Omron HEM-705CP blood pressure monitor at trough (24 hours ± 3 hours post-dose) and recorded at all study visits following detailed directions specified in the study protocol. Three readings were made and msDBP was calculated as the average of the 3 readings. In the event of aberrant readings, ie, the lowest reading was ≥ 10 mmHg systolic or ≥ 5 mmHg diastolic lower than the highest of the 3 readings, 3 additional readings were obtained. A negative change indicates improvement.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Ramipril / Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 61 | 57
mmHg | -6.0 (0.94) | -4.1 (0.96)

4. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study - Aliskiren/Amlodipine vs Ramipril/Amlodipine
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren / Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 60 | 57
mmHg | -5.8 (0.98) | -4.5 (1.00)

5. Secondary Outcome: Percentage of Patients Who Achieved Normalized Blood Pressure at End of Study
Description: Normalized was defined as a msSBP < 140 mmHg and/or a msDBP < 90 mmHg.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 61 | 60 | 57
Percentage of patients | 45.90 | 43.33 | 42.11

6. Secondary Outcome: Change in HOMA-IR From Baseline to End of Study
Description: Homeostasis model assessment-insulin resistance (HOMA-IR) was defined as (fasting insulin [μU/mL] x fasting glucose [mmol/L]) / 22.5.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 45 | 44 | 45
mmol/L | 0.98 (2.292) | 0.87 (5.883) | 0.60 (6.186)

7. Secondary Outcome: Change in HOMA-β From Baseline to End of Study
Description: Homeostasis model assessment-β (HOMA-β) was defined as fasting insulin (μU/mL) x 20 / (fasting glucose (mmol/L) - 3.5).
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 45 | 44 | 45
mmol/L | 2.71 (152.108) | 0.87 (5.883) | 0.60 (6.186)

8. Secondary Outcome: Change in HbA1c (Glycated Hemoglobin) From Baseline to End of Study - Aliskiren/Ramipril/Amlodipine vs Ramipril/Amlodipine
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/mol
Arm/Group | Aliskiren / Ramipril / Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 57 | 54
mmol/mol | 0.1 (0.05) | 0.1 (0.05)

9. Secondary Outcome: Change in HbA1c (Glycated Hemoglobin) From Baseline to End of Study - Aliskiren/Amlodipine vs Ramipril/Amlodipine)
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/mol
Arm/Group | Aliskiren / Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 58 | 54
mmol/mol | 0.1 (0.06) | 0.1 (0.06)

10. Secondary Outcome: Percentage of Patients Who Developed Diabetes at End of Study
Description: A patient had diabetes if fasting plasma glucose > 7 mmol/L.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population: All patients that received at least 1 dose of study drug and had baseline and at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine
Number analyzed (Participants) | 61 | 60 | 57
Percentage of patients | 1.9 | 4.1 | 2.1

ADVERSE EVENTS:
Arm/Group | Aliskiren / Ramipril / Amlodipine | Aliskiren /Amlodipine | Ramipril / Amlodipine
Serious Adverse Events (participants affected / at risk) | 3/61 | 1/60 | 3/57
Other Adverse Events (participants affected / at risk) | 27/61 | 24/60 | 26/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / Ramipril / Amlodipine (N=61) | Aliskiren /Amlodipine (N=60) | Ramipril / Amlodipine (N=57)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Latex allergy (Immune system disorders) | 0 | 1 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0
Glucose tolerance test abnormal (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / Ramipril / Amlodipine (N=61) | Aliskiren /Amlodipine (N=60) | Ramipril / Amlodipine (N=57)
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0
Oedema peripheral (General disorders) | 17 | 14 | 16
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Dizziness (Nervous system disorders) | 5 | 2 | 2
Headache (Nervous system disorders) | 2 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.